CLINICAL TRIAL: NCT04117958
Title: A Global Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of the Half-life Extended Bispecific T-cell Engager AMG 199 in Subjects With MUC17-Positive Solid Tumors Including Gastric, Gastroesophageal Junction, Colorectal, and Pancreatic Cancers
Brief Title: Study of AMG 199 in Subjects With MUC17-Positive Solid Tumors Including Gastric, Gastroesophageal Junction, Colorectal, and Pancreatic Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180290; 2019-002708-42 (EudraCT Number)
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: MUC17-positive Solid Tumors
Keywords: Gastric Cancer; Gastroesophageal Junction Cancer; Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose-exploration phase (Experimental): The dose-exploration phase of the study will estimate the MTD (Maximum Tolerated Dose) of AMG 199 using a Bayesian logistic regression model (BLRM). A RP2D (Recommended Phase 2 Dose) may be identified based on emerging safety, efficacy, and PD (Pharmacodynamics) data prior to reaching an MTD. Alternative dosing schedule(s) may be explored based on emerging PK (Pharmacokinetics) and safety data.
  Interventions: Drug: AMG 199
- Dose-expansion phase (Experimental): The dose-expansion phase will be conducted to confirm safety, PK, and PD at the MTD or RP2D and to obtain further safety and efficacy data and enable correlative biomarker analysis.
  Interventions: Drug: AMG 199

INTERVENTIONS:
Drug: AMG 199 — AMG 199 is a BiTE® molecule designed to direct T cells towards MUC17-expressing cells.

SUMMARY:
To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
AMG 199 is a novel half-life extended (HLE) bispecific T cell engager (BiTE®) molecule designed to direct T cells towards MUC17-expressing cells. This is a first-in-human study in adult subjects with MUC17-positive solid tumors including gastric cancer, gastroesophageal junction (GEJ), colorectal, and pancreatic cancers, collectively referred to as "solid tumors" in this clinical investigation to assess AMG 199 safety, tolerability, pharmacokinetics (PK), and anti-tumor activity, with additional exploratory objectives to assess pharmacodynamics (PD), correlative biomarker analysis, and immunogenicity.

The primary end point is to evaluate the safety and tolerability of AMG 199 in adult subjects, and determine the MTD and RP2D. The secondary end point is characterize the PK and anti-tumor activity of AMG 199.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

• Subjects with histologically or cytologically confirmed metastatic or locally advanced unresectable gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma positive for MUC17. Subjects should have been refractory to or have relapsed after two or more prior lines of standard systemic therapy that included a platinum, a fluoropyrimidine, nivolumab (in combination with a platinum and a fluoropyrimidine), either a taxane or irinotecan, and an approved vascular endothelial growth factor receptor (VEGFR) antibody/tyrosine kinase inhibitor (TKI).

OR

• Subjects with histologically or cytologically confirmed metastatic or locally advanced unresectable colorectal cancer positive for MUC17. Subjects should have been refractory to or have relapsed after at least two and up to five prior lines of standard systemic therapy. Therapy should have included an approved vascular endothelial growth factor (VEGF) antibody (if clinically appropriate) and epidermal growth factor receptor (EGFR) antibody (if kirsten rat sarcoma [KRAS]/ neuroblastoma RAS viral oncogene homolog [NRAS]/ v-Raf murine sarcoma viral oncogene homolog B1 [BRAF] wild type tumor).

OR

* Subjects with histologically or cytologically confirmed unresectable or metastatic pancreatic ductal adenocarcinoma positive for MUC17. Subjects should have been refractory to or have relapsed after at least one and up to three prior lines of standard systemic therapy.
* Gastric adenocarcinoma and GEJ adenocarcinoma: Subjects eligible for human epidermal growth factor receptor 2 (HER2) directed therapy, prior systemic therapy should have an approved HER2 targeting antibody approved for treatment of gastric cancer. For subjects with microsatellite instability high (MSI H) or mismatch repair deficient (dMMR) tumors a prior line of treatment should have included an approved programmed cell death protein-1 (PD-1) blocking antibody.

OR

* Colorectal cancer: For subjects with MSI H or dMMR tumors a prior line of treatment should have included an approved PD-1-blocking antibody. For subjects with BRAF V600E mutation positive tumors a prior line of treatment should have included a BRAF inhibitor.
* Subjects may also be included if the aforementioned therapeutic options were medically not appropriate for them. In these cases, the reason(s) why required prior therapies for solid tumors were medically not appropriate should be documented in the subject's electronic case report form (eCRF). Subjects may also be included if the aforementioned therapeutic options have not been available or accessible for them.
* For dose expansion only: Subjects with at least one measurable lesion ≥ 10mm which has not undergone biopsy within 3 months of screening scan. This lesion cannot be biopsied at any time during the study.

Exclusion Criteria:

Key Exclusion Criteria:

* Any anticancer therapy or immunotherapy within 4 weeks of start of first dose.
* Central nervous system (CNS) metastases, leptomeningeal, or spinal cord compression.
* Autoimmune disorders requiring chronic systemic steroid therapy or any other form of immunosuppressive therapy. Subjects may be included if the treatment is discontinued more than 3 months prior to the first dose of AMG 199, there is a low likelihood of relapse from the autoimmune disorder, AND there is agreement between the investigator and the Amgen Medical Monitor.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicities (DLT) | 3 years
  To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
Incidence of Treatment-emergent adverse events (TEAEs) | 3 years
  To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
Incidence of Treatment-related adverse events (TRAEs) | 3 years
  To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
Number of subjects with changes in vital signs | 3 years
  To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
Number of subjects with changes in clinical laboratory tests | 3 years
  To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
Number of subjects with changes in electrocardiogram (ECG) | 3 years
  To evaluate the safety and tolerability of AMG 199 in adult subjects and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of AMG 199 | 3 years
  To characterize the PK (Pharmacokinetics) of AMG 199.
Minimum serum concentration (Cmin) of AMG 199 | 3 years
  To characterize the PK (Pharmacokinetics) of AMG 199.
Area under the concentration-time curve (AUC) of AMG 199 | 3 years
  To characterize the PK (Pharmacokinetics) of AMG 199.
Accumulation following multiple dosing of AMG 199 | 3 years
  To characterize the PK (Pharmacokinetics) of AMG 199.
Half-life (t1/2) of AMG 199 | 3 years
  To characterize the PK (Pharmacokinetics) of AMG 199.
Objective response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and iRECIST. | 3 years
  To evaluate preliminary anti-tumor activity of AMG 199
Duration of response (DOR). | 3 years
  To evaluate preliminary anti-tumor activity of AMG 199
Time to progression (TTP) | 3 years
  To evaluate preliminary anti-tumor activity of AMG 199
Progression-free survival (PFS), 6-month PFS | 6 months
  To evaluate preliminary anti-tumor activity of AMG 199
Progression-free survival (PFS), 1-year PFS | 1 year
  To evaluate preliminary anti-tumor activity of AMG 199
Overall survival (OS), 1-year OS. | 1 year
  To evaluate preliminary anti-tumor activity of AMG 199
Overall survival (OS), 2-year OS | 2 years
  To evaluate preliminary anti-tumor activity of AMG 199

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - University of California at Irvine Medical Center, Orange, California
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
- Landeskrankenhaus Salzburg, Salzburg, Austria
- Institut Gustave Roussy, Villejuif, France
- Germany (4):
  - Universitaetsklinikum Hamburg Eppendorf Onkologisches Zentrum, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universitaet Muenchen Campus Grosshadern, München
  - Klinikum rechts der Isar, München
- Japan (3):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Netherlands (2):
  - Amsterdam UMC - location VUmc, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com